CLINICAL TRIAL: NCT00355641
Title: A 52-Week, Open-Label Study to Assess the Long-Term Safety of Ropinirole Extended Release (XR) in Patients With Restless Legs Syndrome (RLS)
Brief Title: Long-Term Safety Of Ropinirole XR In Patients With Restless Legs Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101468/206
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Restless Legs Syndrome
Keywords: Ropinirole; Restless Legs Syndrome; RLS
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): All subjects will receive ropinirole XR in this study. The total daily dose range of ropinirole XR will be 0.5mg to 6.0mg daily
  Interventions: Drug: Ropinirole Extended Release (XR)

INTERVENTIONS:
Drug: Ropinirole Extended Release (XR) — Dose range of Ropinirole XR of 0.5mg to 6.0mg daily

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of ropinirole XR in the long-term treatment (up to 52 weeks)of adults with RLS.

ELIGIBILITY:
Inclusion criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Subjects in North America ≥18 years of age who

  1. Have successfully completed one of the following parent studies: 101468/205, ROX104805; OR
  2. Have a diagnosis of primary RLS using the International RLS Study Group (IRSSG) Diagnostic Criteria (Appendix 10), experience RLS symptoms during both the evening (before 8 PM) and night-time, and have a total score ≥15 on the IRLS Rating Scale at Baseline. Subjects must have a history of a minimum of 20 evenings/nights of RLS episodes per month (e.g., any combination of evenings and/or nights for ≥ 20 days). During Screening/Washout, RLS symptoms must be present for at least 4 of 7 evenings/nights immediately prior to the Baseline Visit (e.g., any combination of evenings and/or nights for ≥ 4 days).
* Subjects must give written informed consent prior to any specific study procedures.

Exclusion Criteria:

* Subjects who have any medical conditions which, in the opinion of the investigator, could affect efficacy assessments or clinically significant or unstable medical conditions that present a safety concern. These may include, but are not limited to the following disorders: diabetes, peripheral neuropathy, rheumatoid arthritis, fibromyalgia syndrome, symptomatic orthostatic hypotension, severe cardiovascular disease, hepatic or renal failure, pleuro-pulmonary fibrosis.
* Subjects having clinically significant abnormal laboratory or ECG findings not resolved at time of baseline examinations. Abnormal 12-lead ECG findings include, but are not limited to the following: myocardial ischemia, clinically significant conduction abnormalities, or clinically significant arrhythmias.
* Subjects with a diastolic blood pressure ≥ 110mmHg or ≤ 50mmHg or systolic blood pressure ≥ 180mmHg or ≤ 90mmHg at the Screening or Baseline visit.
* Subjects with a history of augmentation and/or end-of-dose rebound symptoms.

  * Augmentation is defined as RLS symptoms that occurred while on treatment and occur ≥ 2 hours earlier than they did before, symptoms which are more severe than when not treated, symptoms which start after less time at rest than they did before treatment, or symptoms which involve other parts of the body, such as the arms or trunk.
  * End-of-dose rebound is defined as a re-emergence of RLS symptoms in the early morning the day after taking the dose of RLS medication.
* Subjects who have exhibited intolerance to ropinirole.
* For subjects entering Study 206, certain medications must be discontinued prior to entering the study. The following medications are prohibited for the duration of the study period which is up to and including the Follow-up visit:

  ·dopamine agonists (including ropinirole immediate release formulation), dopamine antagonists (e.g., typical neuroleptics, metoclopramide), levodopa/carbidopa The minimum discontinuation period is generally 5 half-lives or 7 consecutive evening/nights medication-free, prior to baseline, whichever is the longer period. If the subject will require longer than 2 weeks following the Follow-up visit of the parent study to complete the washout, GSK must be consulted for further instructions.
* Other medications, including those with partial dopaminergic activity (e.g., atypical antipsychotics, certain antidepressants such as bupropion, tricyclic antidepressants and monoamine oxidase inhibitors) may have additive activity with ropinirole and should be used with caution in patients taking ropinirole. For patients on stable doses, these agents may be permitted; however, it is recommended that the dose of the medication remain stable throughout the duration of the study.
* Night workers or any others whose sleeping habits are incompatible with the study design, or who would be required to make significant changes to their bedtime during the course of the study.
* Women who have a positive pregnancy test.
* Women of child-bearing potential who are not practicing a clinically accepted method of contraception such as oral contraception, surgical sterilization, IUD, diaphragm in conjunction with spermicidal foam and condom on the male partner, or systemic contraception (e.g. Norplant).

The following exclusion criteria must be assessed at Study 206 Screen/Baseline for subjects who are not rolling in following completion of Study 101468/205 or ROX104805:

* Subjects who suffer from a primary sleep disorder other than RLS that may significantly affect the symptoms of RLS (e.g., narcolepsy, sleep terror disorder, sleepwalking disorder, breathing related sleep disorder).
* Subjects diagnosed with movement disorders (e.g., Parkinson's disease, dyskinesias, and dystonias).
* Signs of secondary RLS (e.g., end stage renal disease, iron deficient anemia or pregnancy at Baseline Visit)
* Subjects requiring treatment of daytime RLS symptoms (daytime defined as 7:00 AM until 5:00 PM).
* Subjects with a history of alcohol or substance abuse within the past year.
* Subjects who, in the opinion of the investigator, would be non-compliant with the visit schedule or other study procedures
* Participation in any clinical drug or device trial (other than Study 101468/205 or ROX104805) in the one month prior to the Baseline Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Incidence/severity of adverse events Changes in vital signs Labs ECG Assessment of augmentation and rebound (worsening of RLS symptoms). | Up to 52 Weeks

SECONDARY OUTCOMES:
Change from baseline in IRLS Rating Scale total score CGI Scale scores Medical Outcomes Study Sleep Scale scores Other subject-reported health outcomes. | Up to 52 Weeks
Incidence and severity of adverse events. | Up to 52 Weeks
Changes in vital signs (blood pressure and pulse) and weight. | Up to 52 Weeks
Changes in laboratory assessments (hematology and clinical chemistry). | Up to 52 Weeks
Changes in electrocardiogram (ECG) parameters. | Up to 52 Weeks
Assessment of augmentation. | Up to 52 Weeks
Assessment of rebound. | Up to 52 Weeks
Change from baseline in the IRLS Rating Scale total score at Week 52 LOCF (last observation carried forward). | Up to 52 Weeks
Proportion of subjects with a score of much improved (2) or very much improved (1) on CGI-I at Week 52 LOCF. | Up to 52 Weeks
CGI Severity of Illness (CGI-S) at Week 52 LOCF. | Up to 52 Weeks
Change from baseline in the domains of the Medical Outcomes Study (MOS-12) Sleep Scale at Week 52 LOCF. | Up to 52 Weeks
Change from baseline in the overall life impact score of the RLS Quality of Life Questionnaire at Week 52 LOCF. | Up to 52 Weeks
Change from baseline in the anxiety and depression domains of the Hospital Anxiety and Depression (HADS) Scale at Week 52 LOCF. | Up to 52 Weeks
Change from baseline in the total score and domains of the Profile of Mood States (POMS) Scale Short Form at Week 52 LOCF. | Up to 52 Weeks
Change from baseline in the parameters for the work Productivity and Activity Impairment - Specific Health Problem (WPAI-SHP) Questionnaire at Week 52 LOCF. | Up to 52 Weeks
Proportion of subjects satisfied with their treatment at Week 52 LOCF. | Up to 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (63):
- United States (57):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Reseda, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Dawsonville, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Schenectady, New York
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Canada (6):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] C Hill-Zabala, R Bogan, D Lee, M Lomax. A 52-week open-label study to assess the long-term tolerability of Ropinirole CR Extended Release Tablets in subjects with Restless Legs Syndrome (RLS). 12th International Congress of Parkinson's Disease and Movement Disorders, Chicago, IL, June 22-26, 2008 (abstract 1112).
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 101468/206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101468/206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101468/206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101468/206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 101468/206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101468/206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register